CLINICAL TRIAL: NCT05059795
Title: To Compare the Effectiveness of Various Methods of Estimating Volume Resuscitation in Patients With Cirrhosis With Sepsis Induced Hypotension
Brief Title: Volume Resuscitation in Cirrhosis With Sepsis Induced Hypotension
Status: Completed | Type: Observational
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Madhumita Premkumar, Assitant Professor, Post Graduate Institute of Medical Education and Research, Chandigarh
Other Study IDs: Im/2019/2917
Record Dates: First submitted 2020-07-04; First posted 2021-09-28 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Cirrhosis, Liver; Sepsis; Acute on Chronic Liver Failure
Keywords: Resuscitation in cirrhosis; Inferior vena cava dynamics; Central Venous Pressure in cirrhosis; Lactate clearance in cirrhosis; Acute-on-chronic liver failure; Sepsis in Cirrhosis; Shock in ACLF and Cirrhosis
MeSH Terms: conditions — Liver Cirrhosis; Sepsis; Acute-On-Chronic Liver Failure; Fibrosis | interventions — Albumins; Crystalloid Solutions

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma and Urine Samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Cirrhosis/ACLF of any etiology
  Interventions: Drug: Albumin + electrolyte solution; Diagnostic Test: POCUS guided fluid resuscitation

INTERVENTIONS:
Drug: Albumin + electrolyte solution — Type of resuscitation fluid, dose and use of inotrope
  Other Names: Crystalloid
Diagnostic Test: POCUS guided fluid resuscitation — Conventional goal directed therapy

SUMMARY:
In critically ill patients with liver disease like cirrhosis or ACLF, fluid therapy needs to be instituted after identification of patients who will be fluid responsive and initiate appropriate inotropes early to prevent the mortality associated with fluid overload.

The parameters and methodology used for assessing fluid responsiveness have been studied earlier, but the optimum method is not established. Existing recommendations based on data regarding fluid responsiveness and choice of fluid for resuscitation from intensive care units in general cannot be applied to those with liver disease as the hemodynamic alterations that occur with liver disease, presence of hypoalbuminemia at baseline and presence of cardiac dysfunction interfere with the conventional methods of fluid status assessment, fluid responsiveness as well as the response to different types of resuscitation fluids.

Therefore the investigators attempt to compare various methods to estimate current intravascular volume status of patient which could be helpful in guiding fluid therapy.

DETAILED DESCRIPTION:
Objectives:

1. To compare the accuracy of central venous pressure and inferior vena cava dynamic assessment and lactate clearance for estimating adequacy of fluid resuscitation in patients with cirrhosis with sepsis induced hypotension .[Time Frame at enrolment, 6 hours, 24 hours]
2. Predictors of all-cause mortality at Day 7 and day 28. [Time Frame Day 7 and Day 28]

PATIENTS AND METHODS Study Design: A Prospective observational study

Case Definition:

Cirrhosis will be defined by - "clinical features consistent with chronic liver disease (CLD) including a consistent history as well as a documented complication of CLD (i.e., ascites, varices, hepatic encephalopathy) and/or imaging results consistent with cirrhosis and/or liver histologic findings consistent with cirrhosis" ACLF will be defined as per EASL criteria with documentation of organ failures.

Systemic Inflammatory Response Syndrome (SIRS) - 2 more of following 4

1. Oral temperature >38.3oC or <36oC
2. Heart Rate > 90 beats/min
3. Respiratory Rate >20 breaths/min or PaCO2 <32mmHg
4. WBC count >12000/cumm, <4000/cumm or >10% immature band forms Sepsis is a SIRS in response to proven or suspected microbial event 'Sepsis induced hypotension' implies mean arterial pressure < 65 mmHg or a reduction of >40 mm Hg from baseline in the absence of other causes of hypotension Severe sepsis - sepsis-induced tissue hypoperfusion or organ dysfunction (any of the following thought to be due to the infection)

   * Sepsis-induced hypotension
   * Lactate above upper limits laboratory normal
   * Urine output < 0.5 mL/kg/hr for more than 2 hrs despite adequate fluid resuscitation
   * Acute lung injury with PaO2/FIO2 < 250 in the absence of pneumonia as infection source
   * Acute lung injury with PaO2/FIO2 < 200 in the presence of pneumonia as infection source
   * Creatinine > 2.0 mg/dL (176.8 μmol/L)
   * Bilirubin > 2 mg/dL (34.2 μmol/L)
   * Platelet count < 100,000 μL
   * Coagulopathy (international normalized ratio > 1.5) Septic shock is "sepsis induced hypotension despite adequate fluid resuscitation along with organ dysfunction or perfusion abnormality".

Acute kidney injury (AKI) is defined as any of the following:

1. Increase in SCr by ≥0.3 mg/dl (≥26.5 μmol/l) within 48 hours; or
2. Increase in SCr to ≥1.5 times baseline, which is known or presumed to have occurred within the prior 7 days; or
3. Urine volume <0.5 ml/kg/h for 6 hours

Definition of Adequate Intravascular volume - IVC diameter ≥ 18mm and IVCCI <40% Definition of Adequate fluid resuscitation - Achieving MAP ≥ 65mmHg with Fluid bolus

All patients eligible for the study will undergo screening as per the above criteria. The ones who satisfy the criteria will be counselled for participation in the study and written informed consent will be taken from the patient / the legal guardian in patients who are unable to do so. Patient information sheets will also be signed, briefing the patients about why the research work is necessary and also about the methodology.

Detail history and clinical examination will be done in all cases and the findings along with all investigation results will be recorded in a standard case record form. Information would be collected regarding the onset and duration of symptoms, etiology, and severity of disease, other baseline clinical features, demographic characteristics, routine biochemical and hematological investigations.

* After enrolment, baseline samples would be taken for routine investigations and samples for evaluation of sepsis - blood culture, urine culture, fluid cultures, procalcitonin will be taken.
* The patient would be assessed for 5 parameters and will be reassessed 30min and 4hours after starting fluid resuscitation.

  1. IVC diameter and collapsibility Index
  2. Serum lactate levels
  3. Venous-arterial pCO2 difference
  4. CVP where central line inserted as per treating physician's decision
  5. ScVO2 where central line available
* The patients in septic shock where IVC diameter <18mm or IVCCI≥40% in spontaneously breathing patients, would be regarded in fluid depleted state and will be given aggressive fluid resuscitation with 20% albumin 100 ml started within 30 min which is a standard fluid of choice in patients with cirrhosis and other fluids - Normal Saline/ balanced salt solution 30ml/kg over 3hrs.

(The patients who not fulfil above criteria would be assumed in a fluid replete state and be started on maintenance fluid management along with inotrope support as per standard dosage guidelines) Norepinephrine would be 1st choice vasopressor - started at a dose of 4μg/min and titrated every 20 min to a maximum of 21.3μg/min. If MAP still <65mmHg, Vasopressor would be added starting from a 0.01U/min to 0.04U/min. Adrenaline would be added in shock refractory to both vasopressors in dose of 4-24μg/min.

* Along with fluid and inotrope support, the patient will also receive standard of care including empiric broad spectrum antibiotics, oxygen support/ventilator support if needed.
* MAP would be rechecked 30 min after starting fluid therapy. IVC diameter and IVCCI would also be checked at same time to see if change in MAP (if any) is reflected in the IVC status. Adequate fluid resuscitation would be defined by achieving a MAP ≥ 65mmHg. In patients achieving MAP≥65mmHg, fluid therapy will be continued. The patients still having MAP<65 mmHg will be started on inotrope support according to standard guidelines.
* IVC, IVCCI, Lactate, venous-arterial pCO2 difference, CVP and ScVO2 would be remeasured at 4 hrs.
* The patient would be the followed with serial examinations, calculations of SOFA score, CTP and MELD.
* Samples to test for sepsis such as procalcitonin, galactomannan, beta D Glucan and high sensitivity CRP will be done every 48-72 hours as determined by the treating clinician.
* Cultures for bacterial and fungal sepsis will be taken as per the Liver ICU protocol.
* If discharged earlier, for the purpose of 28-day mortality the patients' kin would be contacted telephonically.
* Data regarding total amount of fluids, type of fluids, urine output, dose and duration of inotropes, initiation of RRT, total days in ICU/Hospital, immediate cause of death (In case of mortality) would be noted.

Presence of Cirrhotic Cardiomyopathy as per updated 2020 CCMC criteria.

CCM is defined as systolic or diastolic dysfunction in the absence of alternative cardiac pathology in concordance with the Cirrhotic Cardiomyopathy Consortium (CCMC) criteria. 9 Systolic dysfunction was defined as an ejection fraction (EF) ≤50% or an absolute value of GLS <18%. LVDD will be defined as presence of 3 of the following 4 criteria: septal early diastolic mitral annular flow velocity (e') <7 cm/s, early diastolic transmitral flow to early diastolic mitral annular velocity (E/e') ≥15, left atrial volume index (LAVI) >34 mL/m2, tricuspid jet maximum velocity >2.8 m/s, in the absence of pulmonary hypertension and the presence of measurable early to late diastolic transmitral flow velocity (E/A) ratio (E/A >2 = grade 3 & E/A 0.8-2 = grade 2 LVDD). Persons meeting only 2 criteria will be termed as indeterminate for LVDD grade. 19

ELIGIBILITY:
Inclusion Criteria:

1. Clinical/Imaging or Biopsy proven liver cirrhosis of any etiology
2. Hypotension (MAP <65mmHg or SBP <90mmHg)
3. 18-65 yrs of age

Exclusion Criteria:

1. Already received colloid or 2 litres of fluid within the first 2 hours of presentation, without echocardiographic assessment.
2. Already on vasopressors/inotropes
3. Severe pre-existing cardiopulmonary disease
4. Acute Respiratory Distress Syndrome (ARDS)
5. Active bleeding like variceal bleed 28
6. Cerebrovascular events
7. Chronic renal disease - End Stage Renal Disease (ESRD)/ patient on renal replacement therapy
8. Admission to ICU following liver transplantation, burns, cardiac surgery
9. Brain death or likely brain death within 24 hours
10. Previous adverse reaction to human albumin solution
11. Pregnant or lactating women
12. Informed consent refused by patient or attendants

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients 18-65 years age with cirrhosis of any etiology now presenting with sepsis induced hypotension
Sampling Method: Probability Sample
Enrollment: 350 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-08-10 (Actual)

PRIMARY OUTCOMES:
Achievement of Mean Arterial pressure >65 mmHg | At the end of 4 hours since admission (time zero)

SECONDARY OUTCOMES:
Requirement of vasopressors | At the end of 4 hours of admission
Requirement of vasopressors | At the end of 24 hours of admission
Volume of fluid infused | At the end of 4 hours of admission
  Dose of albumin
Volume of fluid infused | At the end of 24 hours of admission
  Dose of crystalloid
Volume of fluid infused | At the end of 36 hours of admission
  Total volume of fluids
Volume of fluid infused | At the end of 48 hours of admission
  Dose of albumin and crystalloid
Volume of fluid infused | At the end of 72 hours of admission
  Dose of albumin and crystalloid
Incidence of Acute Kidney Injury | At admission
Incidence of Acute Kidney Injury | Day 7
  Any new episode of AKI documented in the first week of admission
Incidence of new organ dysfunction (encephalopathy, coagulation failure, respiratory failure) | Day 7
  Any new episode of new organ dysfunction documented in the first week of admission
Duration of ICU stay | Total duration of ICU stay in days
  The total duration of stay in intensive care, which will be assessed till 28 days
Duration of hospital stay | Total duration of admission as a hospital inpatient, assessed till 28 days
  The total duration of stay in hospital, which will be assessed till 28 days
Mortality | Day 7
  Incidence of death at the end of 1 week i.e. early mortality
Mortality | Day 28
  Incidence of death at the end of 4 weeks i.e. late mortality
Documentation of Cardiac index | Time zero at admission
  POC ultrasound and echocardiography documentation (Cardiac index), Systemic Vascular resistance index (SVRI) 0h,6h on day 1
Documentation of Cardiac index at 6h | At 6 hours of admission
  POC ultrasound and echocardiography documentation (Cardiac index), Systemic Vascular resistance index (SVRI) 0h,6h on day 1
Documentation of Cardiac index at 24h | At 24 hours of admission
  POC ultrasound and echocardiography documentation (Cardiac index), Systemic Vascular resistance index (SVRI) 0h,6h on day 1
Documentation of Cardiac index at 48h | At 48 hours of admission
  POC ultrasound and echocardiography documentation (Cardiac index), Systemic Vascular resistance index (SVRI) 0h,6h on day 1
Documentation of Cardiac index at 72h | At 72 hours of admission
  POC ultrasound and echocardiography documentation (Cardiac index), Systemic Vascular resistance index (SVRI) 0h,6h on day 1
Documentation of POCUS systemic vascular resistance index | Time zero at admission
  POC ultrasound and echocardiography documentation for changes in (Cardiac index), Systemic Vascular resistance index (SVRI)
Documentation of POCUS systemic vascular resistance index at 6h | at 6hours of admission
  POC ultrasound and echocardiography documentation for changes in (Cardiac index), Systemic Vascular resistance index (SVRI)
Documentation of POCUS systemic vascular resistance index at 24h | at 24hours of admission
  POC ultrasound and echocardiography documentation for changes in (Cardiac index), Systemic Vascular resistance index (SVRI)
Documentation of POCUS systemic vascular resistance index at 48h | at 48hours of admission
  POC ultrasound and echocardiography documentation for changes in (Cardiac index), Systemic Vascular resistance index (SVRI)
Documentation of POCUS systemic vascular resistance index at 72h | at 72hours of admission
  POC ultrasound and echocardiography documentation for changes in (Cardiac index), Systemic Vascular resistance index (SVRI)
Documentation of IVC dynamics | time zero at admission (Day 0)
  POC ultrasound and echocardiography documentation for changes in (Cardiac index), Systemic Vascular resistance index (SVRI)
Documentation of IVC dynamics | At 6hours of admission (Day 1)
  POC ultrasound and echocardiography documentation for changes in (Cardiac index), Systemic Vascular resistance index (SVRI)
Documentation of IVC dynamics | at 24hours of admission
  POC ultrasound and echocardiography documentation for changes in echo parameters (Cardiac index), Systemic Vascular resistance index (SVRI)
Documentation of IVC dynamics | at 48hours of admission
  POC ultrasound and echocardiography documentation for changes in echo parameters (Cardiac index), Systemic Vascular resistance index (SVRI)
Documentation of IVC dynamics | at 72hours of admission
  POC ultrasound and echocardiography documentation for changes in echo parameters (Cardiac index), Systemic Vascular resistance index (SVRI)

CONTACTS AND LOCATIONS:
Locations (2):
- India (2):
  - PGIMER, Chandigarh, Chandigarh
  - Postgraduate Institute of Medical Education and Research, Chandigarh

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Moreau R, Hadengue A, Soupison T, Kirstetter P, Mamzer MF, Vanjak D, Vauquelin P, Assous M, Sicot C. Septic shock in patients with cirrhosis: hemodynamic and metabolic characteristics and intensive care unit outcome. Crit Care Med. 1992 Jun;20(6):746-50. doi: 10.1097/00003246-199206000-00008. PMID 1597026
- [Background] ARISE Investigators; ANZICS Clinical Trials Group; Peake SL, Delaney A, Bailey M, Bellomo R, Cameron PA, Cooper DJ, Higgins AM, Holdgate A, Howe BD, Webb SA, Williams P. Goal-directed resuscitation for patients with early septic shock. N Engl J Med. 2014 Oct 16;371(16):1496-506. doi: 10.1056/NEJMoa1404380. Epub 2014 Oct 1. PMID 25272316
- [Background] Marik PE, Baram M, Vahid B. Does central venous pressure predict fluid responsiveness? A systematic review of the literature and the tale of seven mares. Chest. 2008 Jul;134(1):172-8. doi: 10.1378/chest.07-2331. PMID 18628220
- [Background] Bentzer P, Griesdale DE, Boyd J, MacLean K, Sirounis D, Ayas NT. Will This Hemodynamically Unstable Patient Respond to a Bolus of Intravenous Fluids? JAMA. 2016 Sep 27;316(12):1298-309. doi: 10.1001/jama.2016.12310. PMID 27673307
- [Background] Velissaris D, Pierrakos C, Scolletta S, De Backer D, Vincent JL. High mixed venous oxygen saturation levels do not exclude fluid responsiveness in critically ill septic patients. Crit Care. 2011 Jul 26;15(4):R177. doi: 10.1186/cc10326. PMID 21791090
- [Background] Lee YK, Hwang SY, Shin TG, Jo IJ, Suh GY, Jeon K. Prognostic Value of Lactate and Central Venous Oxygen Saturation after Early Resuscitation in Sepsis Patients. PLoS One. 2016 Apr 7;11(4):e0153305. doi: 10.1371/journal.pone.0153305. eCollection 2016. PMID 27054713
- [Background] Lee J, de Louw E, Niemi M, Nelson R, Mark RG, Celi LA, Mukamal KJ, Danziger J. Association between fluid balance and survival in critically ill patients. J Intern Med. 2015 Apr;277(4):468-77. doi: 10.1111/joim.12274. Epub 2014 Jun 27. PMID 24931482
- [Background] Sefidbakht S, Assadsangabi R, Abbasi HR, Nabavizadeh A. Sonographic measurement of the inferior vena cava as a predictor of shock in trauma patients. Emerg Radiol. 2007 Jul;14(3):181-5. doi: 10.1007/s10140-007-0602-4. Epub 2007 Jun 1. PMID 17541661
- [Background] Premkumar M, Rangegowda D, Kajal K, Khumuckham JS. Noninvasive estimation of intravascular volume status in cirrhosis by dynamic size and collapsibility indices of the inferior vena cava using bedside echocardiography. JGH Open. 2019 Mar 12;3(4):322-328. doi: 10.1002/jgh3.12166. eCollection 2019 Aug. PMID 31406926
- [Background] Jansen TC, van Bommel J, Schoonderbeek FJ, Sleeswijk Visser SJ, van der Klooster JM, Lima AP, Willemsen SP, Bakker J; LACTATE study group. Early lactate-guided therapy in intensive care unit patients: a multicenter, open-label, randomized controlled trial. Am J Respir Crit Care Med. 2010 Sep 15;182(6):752-61. doi: 10.1164/rccm.200912-1918OC. Epub 2010 May 12. PMID 20463176
- [Background] Du W, Liu DW, Wang XT, Long Y, Chai WZ, Zhou X, Rui X. Combining central venous-to-arterial partial pressure of carbon dioxide difference and central venous oxygen saturation to guide resuscitation in septic shock. J Crit Care. 2013 Dec;28(6):1110.e1-5. doi: 10.1016/j.jcrc.2013.07.049. PMID 24216336
- [Background] Izzy M, VanWagner LB, Lin G, Altieri M, Findlay JY, Oh JK, Watt KD, Lee SS; Cirrhotic Cardiomyopathy Consortium. Redefining Cirrhotic Cardiomyopathy for the Modern Era. Hepatology. 2020 Jan;71(1):334-345. doi: 10.1002/hep.30875. Epub 2019 Oct 11. PMID 31342529